CLINICAL TRIAL: NCT01209676
Title: A Phase 0, Exploratory Study of the Pharmacodynamics of a Single Intratumoral Dose of IMCgp100, a Monoclonal Receptor Anti-CD3 scFv Fusion Protein, in Subjects With Advanced Unresectable Melanoma
Brief Title: IMCgp100 in Advanced Unresectable Melanoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 03610
Record Dates: First submitted 2010-09-22; First posted 2010-09-27 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Melanoma; Advanced Disease; Unresectable
Keywords: melanoma, with advanced unresectable
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMCgp100 (Experimental): IMCgp100 will be injected cutaneously or subcutaneously into the metastasis, and peritumoral area if applicable
  Interventions: Drug: IMCgp100 injection

INTERVENTIONS:
Drug: IMCgp100 injection — a monoclonal T cell receptor anti-CD3scFv fusion protein

SUMMARY:
A phase 0, exploratory study of the pharmacodynamics of a single intratumoral dose of IMCgp100, a monoclonal T cell receptor anti-CD3 scFv fusion protein, in subjects with advanced unresectable melanoma to assess the safety and pharmacodynamic properties of single intratumoral doses of IMCgp100 in the setting of advanced unresectable melanoma. Six patients will be enrolled to complete the study over approximately 12-15 months.

DETAILED DESCRIPTION:
This study will test the safety effect of a single dose of the investigational drug IMCgp100 when administered directly into the metastatic melanoma lesion in patients with advanced metastatic melanoma. IMCgp100 is a drug made up of two components. The first is the T cell receptor designed to bind specifically and tightly with protein found at high levels on the surface of melanoma cancer cells and second is an anti-CD3 fragment that is meant to bind to and activate the T cells. There will be two stage dose regimens each enrolling 3 patients. Stage 1 dose will 0.00017 mg IMCgp100 and Stage 2 dose will be 0.0017 mg IMCgp100. Inclusion Criteria: 1. Histologically confirmed dx of advanced unresectable melanoma not requiring immediate treatment and/or in a window between treatments 2. Two or more cutaneous or subcutaneous melanoma metastatic lesions 7 to 15 mm in at least one dimension and amenable to subsequent biopsy 3. Greater or equal to 18 years of age 4. ECOG PS 0-2 5.

Able to provide informed consent and willing to comply with protocol requirements 6. Female patients must not be of childbearing potential or must have negative serum pregnancy test 48 hours prior to receiving investigational drug 7. Male patients must agree to use reliable form of birth control throughout study 8. Must have adequate organ system function Exclusion Criteria: 1. Received any other chemo, immune, radiation or investigational therapy agents within 2 weeks prior to study treatment 2. Cutaneous metastasis that have received prior local therapy 3. Pregnant or breastfeeding 4.

History of autoimmune disease 5. Current treatment with steroid or other immunosuppressive meds 6. Active uncontrolled infection 7. Known HIV infection 8. Uncontrolled seizures 9. Known delayed wound healing 10. On full dose anticoagulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed diagnosis of melanoma, with advanced unresectable disease not currently requiring immediate treatment and/or in a window between treatments.
* 2. Two or more cutaneous or subcutaneous melanoma metastatic lesions 7-15 mm in at least one dimension and amenable to subsequent biopsy.
* 3. Age 18 years
* 4. ECOG performance status 0-2
* 5. Able to understand and to provide written informed consent and willingness to comply with all protocol requirements;
* 6. Female patients who are not be of childbearing potential as documented by medical history (e.g., tubal ligation or hysterectomy), or be post menopausal with a minimum 1 year without menses or have a negative serum beta human chorionic gonadotropin (HGC) pregnancy test within 48 hours prior to receiving the intratumoral injection and agree to use an acceptable form of birth control, defined as abstinence or use of an intrauterine device (IUD), oral contraceptive, barrier and spermicide, or hormonal implant throughout the study period;
* 7. Male patients who must agree to use an acceptable form of birth control throughout the study period.
* 8. Adequate organ system function as evidenced by laboratory values: -Absolute neutrophil count (ANC) greater than or equal to 1.0 X 109/L -Hemoglobin greater than or equal to 9 g/dL -Platelets greater than or equal to 75 X 109/L -Total bilirubin less than or equal to 1.5 mg/dL -AST and ALT less than or equal to 2.5 X ULN ( 2.5 X ULN in the presence of liver metastasis.) -Creatinine less than or equal to 2 mg/dL -TSH within normal limits -INR/PT and PTT less than or equal to 1.3 X ULN

Exclusion Criteria:

* 1. Receive any chemotherapy, immunotherapy, radiation therapy, or other investigational agents (agents part of a research protocol or not approved by the FDA) within 2 weeks prior to injection. A minimum of 14 days is required between last therapy and injection on this study. In addition, any clinically significant drug-related toxicity should have recovered to grade 1 or less (excluding alopecia)
* 2. Patients without cutaneous or subcutaneous metastatic lesions;
* 3. Cutaneous metastases that have received prior local therapy, such as radiation or isolated limb perfusion.
* 4. Pregnancy or breastfeeding
* 5. History of autoimmune disease (excluding vitiligo or controlled thyroid disease) or immunodeficiency.
* 6. Current treatment with steroids (inhaled, topical or systemic) or other immunosuppressive medications within 2 weeks of injection;
* 7. Active uncontrolled infection;
* 8. Known HIV positivity;
* 9. Uncontrollable seizures;
* 10. Known delayed wound healing;
* 11. Full dose anticoagulation with heparin, warfarin, or any other anticoagulant within 2 weeks of injection ;
* 12. History of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting, stroke or TIA within the past 24 weeks.;
* 13. Known hypersensitivity of IMCgp100 or any of its components (ie, Tween) ;
* 14. Class II, III, or IV heart failure as defined by the New York Heart Association;
* 15. Any psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* 16. Any other condition that in the investigators opinion would jeopardize compliance with the protocol ;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Adverse Events as a Measure of Safety and Tolerability | 15 months
  To determine the safety and pharmacodynamic properties of single intratumoral doses of IMCgp100 in the setting of advanced unresectable melanoma.
  Tumor Lesions, peripheral blood pre- and post-injection will be used to determine the safety and pharmacodynamic properties of single intratumoral doses of IMCgp100 in the setting of advanced unresectable melanoma

SECONDARY OUTCOMES:
Adverse events | 15 months
  Will be used to determine the safety and tolerability of IMCgp100 at subtherapeutic doses.
Vital signs | 15 months
  will be used to determine the safety and tolerability of IMCgp100 at subtherapeutic doses.
PE examinations findings | 15 months
  will be used to determine the safety and tolerability of IMCgp 100 at subtherapeutic doses.
Peripheral blood samples | 15 months
  will be used to examine peripheral cytokine measurements as evidence of product immunoactivity and peripheral T and NK cell numbers, phenotype and activation marker status.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgos Karakousis, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States